CLINICAL TRIAL: NCT01998958
Title: A Double-Blind, Doubly-Randomized, Placebo-Controlled Study of Intranasal Esketamine in an Adaptive Treatment Protocol to Assess Safety and Efficacy in Treatment-Resistant Depression (SYNAPSE)
Brief Title: A Study to Evaluate the Safety and Efficacy of Intranasal Esketamine in Treatment-resistant Depression
Acronym: SYNAPSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR102968; 2013-004005-11 (EudraCT Number); JNJ-54135419 (Other: Janssen Research & Development, LLC); ESKETINTRD2003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Results first posted 2019-06-12 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Treatment Resistant Depressive Disorder
Keywords: Treatment resistant depressive disorder; Intranasal esketamine; Efficacy; SYNAPSE; JNJ-54135419
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (5):
- Esketamine 14 mg (Experimental): Participants in Panel B will self-administer intranasal esketamine 14 milligram or placebo on Days 1, 4, 8, and 11 during the double-blind phase and intranasal esketamine on Days 15, 18, 22, and 25 during the optional open-label phase. During the optional open-label phase, participants will start with treatment with a 56-mg dose of intranasal esketamine on Day 15 (the dose of esketamine can be adjusted if desired based on the Investigator's clinical judgment of efficacy and tolerability).
  Interventions: Drug: Esketamine 14 mg; Drug: Esketamine 56 mg; Drug: Placebo
- Esketamine 28 mg (Experimental): Participants in Panel A will self-administer intranasal esketamine 28 mg or placebo on Days 1, 4, 8, and 11 during the double-blind phase and intranasal esketamine on Days 15, 18, 22, 25, 32, 39, 46, 60, and 74 during the optional open-label phase. During the optional open-label phase, all participants will start treatment with a 56-mg dose of intranasal esketamine on Day 15 (the dose of esketamine can be adjusted if desired based on the Investigator's clinical judgment of efficacy and tolerability).
  Interventions: Drug: Esketamine 28 mg; Drug: Esketamine 56 mg; Drug: Placebo
- Esketamine 56 mg (Experimental): Participants in Panel A and Panel B will self-administer intranasal esketamine 56 mg or placebo on Days 1, 4, 8, and 11 during the double-blind phase. During the optional open-label phase, participants in Panel A will self-administer intranasal esketamine on Days 15, 18, 22, 25, 32, 39, 46, 60, and 74 and participants in Panel B will self-administer intranasal esketamine on Days 15, 18, 22, and 25. During the optional open-label phase, all participants will start treatment with a 56-mg dose of intranasal esketamine on Day 15 (the dose of esketamine can be adjusted if desired based on the Investigator's clinical judgment of efficacy and tolerability).
  Interventions: Drug: Esketamine 56 mg; Drug: Placebo
- Esketamine 84 mg (Experimental): Participants in Panel A will self-administer intranasal esketamine 84 mg or placebo on Days 1, 4, 8, and 11 during the double-blind phase and intranasal esketamine on Days 15, 18, 22, 25, 32, 39, 46, 60, and 74 during the optional open-label phase. During the optional open-label phase, all participants will start treatment with a 56-mg dose of intranasal esketamine on Day 15 (the dose of esketamine can be adjusted if desired based on the Investigator's clinical judgment of efficacy and tolerability).
  Interventions: Drug: Esketamine 56 mg; Drug: Esketamine 84 mg; Drug: Placebo
- Placebo (Placebo Comparator): Participants in Panel A and B will self-administer intranasal placebo on Days 1 and 4 during the double-blind phase. Depending on response on Day 8, participants will receive intranasal placebo on Days 8 and 11 or be re-randomized to receive intranasal placebo or esketamine at a dose of 28 mg, 56 mg, or 84 mg (Panel A) or 14 mg or 56 mg (Panel B) on Day 8 and Day 11.
  Interventions: Drug: Esketamine 14 mg; Drug: Esketamine 28 mg; Drug: Esketamine 56 mg; Drug: Esketamine 84 mg; Drug: Placebo

INTERVENTIONS:
Drug: Esketamine 14 mg — 1 to 6 sprays of esketamine 14 mg self-administered as an intranasal formulation for 4 days (Days 1, 4, 8, 11) during the double-blind phase and if applicable during the optional open-label phase for up to 4 days
  Arms: Esketamine 14 mg; Placebo
Drug: Esketamine 28 mg — 1 to 6 sprays of esketamine 28 mg self-administered as an intranasal formulation for 4 days (Days 1,4, 8, 11) during the double-blind phase and if applicable, during the optional open-label phase for up to 9 days
  Arms: Esketamine 28 mg; Placebo
Drug: Esketamine 56 mg — 1 to 6 sprays of esketamine 56 mg self-administered as an intranasal formulation for up to 4 days (Days 1, 4, 8, 11) during the double-blind phase and if applicable, during the optional open-label phase for up to 9 days
Drug: Esketamine 84 mg — 1 to 6 sprays of esketamine 84 mg self-administered as an intranasal formulation for up to 4 days (Days 1, 4, 8, 11) during the double-blind phase and if applicable, during the optional open-label phase for up to 9 days
  Arms: Esketamine 84 mg; Placebo
Drug: Placebo — 1 to 6 sprays of placebo self-administered as an intranasal formulation for 2 days (Days 1 and 4) or depending on response on Day 8, for 4 days (Days 1,4, 8, 11) during the double-blind phase

SUMMARY:
The purpose of this study is to assess the efficacy and dose response of intranasal esketamine (Panel A: 28 mg, 56 mg, and 84 mg and Panel B: 14 mg and 56 mg) compared with placebo in improving depressive symptoms in participants with treatment-resistant depression (TRD).

DETAILED DESCRIPTION:
This will be a 2-panel, randomized ( participants are assigned different treatments based on chance), double-blind (neither investigator nor participant knows which treatment the participant receives), placebo-controlled (placebo is an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial), multicenter study. Approximately 100 male and female adult participants diagnosed with TRD will participate in this study. For participants in both panels (Panel A and Panel B), there will be 4 study phases: a 4-week screening phase, a double-blind treatment phase (Day 1 to Day 15), an optional open-label treatment phase (Panel A: Day 15 to 74; Panel B: Day 15 to 25), and an 8-week post-treatment (follow-up) phase. Depending on the treatment Panel, patients will be assigned to intranasal placebo or intranasal esketamine 14 mg, 28 mg, 56 mg, or 84 mg. Safety assessments will be performed throughout the study. The maximum study duration for a participant will be 23 weeks for Panel A and 16 weeks for Panel B.

ELIGIBILITY:
Inclusion Criteria:

--Participant must meet Diagnostic and Statistical Manual of Mental Disorders -Fourth Edition -Text Revised (DSM-IV-TR) diagnostic criteria for Major Depressive Disorder (MDD), without psychotic features, based upon clinical assessment, and confirmed by the Mini International Neuropsychiatric Interview (MINI)-Participant's major depressive episode and treatment response must be deemed "valid" by remote independent raters-Participant must have had an inadequate response to at least 2 antidepressants, at least one of which is in the current episode of depression; the antidepressant treatment response questionnaire (ATRQ) will be used to assess antidepressant treatment response during the current episode; prior medication history will be used to determine antidepressant treatment response in prior episode(s) -Have an Inventory of Depressive Symptoms-Clinician rated, 30-item (IDS-C30) total score >=34 at Screening and predose at Day 1

Exclusion Criteria:

-Participant has a current DSM-IV-TR diagnosis of bipolar and related disorders, intellectual disability, or cluster b personality disorder (e.g., borderline personality disorder, antisocial personality disorder, histrionic personality disorder, and narcissistic personality disorder) -Participant has a current or prior DSM-IV-TR diagnosis of a psychotic disorder, MDD with psychosis, post-traumatic stress disorder (PTSD), or obsessive compulsive disorder (OCD) -Anatomical or medical conditions that may impede delivery or absorption of study medication (e.g., undergone facial reconstruction, rhinoplasty, significant structural or functional abnormalities of the nose or upper airway; obstructions or mucosal lesions of the nostrils or nasal passages; undergone sinus surgery in the previous 2 years; signs and symptoms of rhinitis) -Has an abnormal or deviated nasal septum with any 1 or more of the following symptoms: blockage of 1 or both nostrils, nasal congestion (especially 1-sided), frequent nosebleeds, frequent sinus infections, and at times has facial pain, headaches, and postnasal drip -Has a history of substance abuse (drug or alcohol) or dependence (except nicotine or caffeine) within the previous 1 year of the screening visit -Participant has known allergies, hypersensitivity, intolerance, or contraindication to esketamine/ketamine or its excipients

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2014-01-27 (Actual); Primary Completion 2015-07-21 (Actual); Study Completion 2015-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (25):
- United States (14):
  - Birmingham, Alabama
  - Garden Grove, California
  - Hartford, Connecticut
  - Jacksonville, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Rockville, Maryland
  - Cedarhurst, New York
  - New York, New York
  - Allentown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
- Lede, Belgium
- Japan (10):
  - Akita
  - Hiroshima
  - Ichikawa
  - Kanzaki
  - Kashihara
  - Kitakyushu
  - Kodaira
  - Kumamoto
  - Nagano
  - Shibukawa

REFERENCES:
- [Derived] Perez-Ruixo C, Rossenu S, Zannikos P, Nandy P, Singh J, Drevets WC, Perez-Ruixo JJ. Population Pharmacokinetics of Esketamine Nasal Spray and its Metabolite Noresketamine in Healthy Subjects and Patients with Treatment-Resistant Depression. Clin Pharmacokinet. 2021 Apr;60(4):501-516. doi: 10.1007/s40262-020-00953-4. Epub 2020 Oct 31. PMID 33128208
- [Derived] Daly EJ, Singh JB, Fedgchin M, Cooper K, Lim P, Shelton RC, Thase ME, Winokur A, Van Nueten L, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine Adjunctive to Oral Antidepressant Therapy in Treatment-Resistant Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Feb 1;75(2):139-148. doi: 10.1001/jamapsychiatry.2017.3739. PMID 29282469
- See also: A Double-Blind, Doubly-Randomized, Placebo-Controlled Study of Intranasal Esketamine in an Adaptive Treatment Protocol to Assess Safety and Efficacy in Treatment-Resistant Depression — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR102968&attachmentIdentifier=71cc4b21-a4b5-44af-8c9b-04d0131f96f4&fileName=ESKETINTRD2003_(CR102968)_Additional_results_data_CH.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Panel A: Period 1): Participants self-administered placebo intranasally (1 spray to each nostril at 0, 5 and 10 minutes) on Days 1 and 4 of Period 1 in Panel A.
- Esketamine 28 mg (Panel A: Period 1): Participants self administered esketamine 28 milligram (mg) intranasally (1 spray of esketamine 14 mg to each nostril at 0 minute and 1 spray of placebo to each nostril at 5 and 10 minutes) on Days 1 and 4 of Period 1 in Panel A.
- Esketamine 56 mg (Panel A: Period 1): Participants self administered esketamine 56 mg intranasally (1 spray of esketamine 14 mg to each nostril at 0 and 5 minute and 1 spray of placebo to each nostril at 10 minutes) on Days 1 and 4 of Period 1 in Panel A.
- Esketamine 84 mg (Panel A: Period 1): Participants self administered esketamine 84 mg intranasally (1 spray of esketamine 14 mg to each nostril at 0, 5 and 10 minutes) on Days 1 and 4 of Period 1 in Panel A.
- Placebo (Panel B: Period 1): Participants self administered placebo intranasally (1 spray to each nostril at 0 and 5 minutes) on Days 1 and 4 of Period 1 in Panel B.
- Esketamine 14 mg (Panel B: Period 1): Participants self administered esketamine 14 mg intranasally (1 spray of esketamine 14 mg into one nostril and 1 spray of placebo into other nostril at 0 minute and then 1 spray of placebo to each nostril at 5 minutes) on Days 1 and 4 of Period 1 in Panel B.
- Esketamine 56 mg (Panel B: Period 1): Participants self administered esketamine 56 mg intranasally (1 spray of esketamine 14 mg into each nostril at 0 and 5 minutes) on Days 1 and 4 of Period 1 in Panel B.
- Placebo (Panel A: Period 2) QIDS >= 11 Participants: Participants who were non-responders at the end of Period 1 in Panel A (with QIDS-SR16 score greater than or equal to [>=] 11) were re-randomized to receive Placebo (1 spray to each nostril at 0, 5 and 10 minutes) on Days 8 and 11 of Period 2.
- Placebo (Panel A: Period 2) QIDS<11 Participants: Participants who were responders (with QIDS-SR16 score <11) at the end of Period 1 in Panel A continued to receive placebo (1 spray to each nostril at 0, 5 and 10 minutes) on Days 8 and 11 of Period 2.
- Placebo to Esketamine 28mg (Panel A: Period 2): Participants who were non-responders at the end of Period 1 in Panel A (with QIDS-SR16 score >=11) were re-randomized to receive esketamine 28 mg (1 spray of esketamine 14 mg to each nostril at 0 minute and 1 spray of placebo to each nostril at 5 and 10 minutes) on Days 8 and 11 of Period 2.
- Placebo to Esketamine 56 mg (Panel A: Period 2): Participants who were non-responders at the end of Period 1 in Panel A (with QIDS-SR16 score >=11) were re-randomized to receive esketamine 56 mg (1 spray of esketamine 14 mg to each nostril at 0 and 5 minute and 1 spray of placebo to each nostril at 10 minutes) on Days 8 and 11 of Period 2.
- Placebo to Esketamine 84 mg (Panel A: Period 2): Participants who were non-responders at the end of Period 1 in Panel A (with QIDS-SR16 score >=11) were re-randomized to receive esketamine 84 mg (1 spray of esketamine 14 mg to each nostril at 0, 5 and 10 minutes) on Days 8 and 11 of Period 2.
- Esketamine 28 mg (Panel A: Period 2): Participants who received esketamine 28 mg in Period 1 of Panel A continued to receive esketamine 28 mg (1 spray of esketamine 14 mg to each nostril at 0 minute and 1 spray of placebo to each nostril at 5 and 10 minutes) on Days 8 and 11 of Period 2.
- Esketamine 56 mg (Panel A: Period 2): Participants who received esketamine 56 mg in Period 1 of Panel A continued to receive esketamine 56 mg (1 spray of esketamine 14 mg to each nostril at 0 and 5 minute and 1 spray of placebo to each nostril at 10 minutes) on Days 8 and 11 of Period 2.
- Esketamine 84 mg (Panel A: Period 2): Participants who received esketamine 84 mg in Period 1 of Panel A continued to receive esketamine 84 mg (1 spray of esketamine 14 mg to each nostril at 0, 5 and 10 minutes) on Days 8 and 11 of Period 2.
- Placebo (Panel B: Period 2) QIDS >=11 Participants: Participants who were non-responders with QIDS-SR16 score >=11 at the end of Period 1 were re-randomized to receive placebo intranasally (1 spray of placebo into each nostril at 0 and 5 minutes using 4 separate devices) on Days 8 and 11 of Period 2 in Panel B.
- Placebo (Panel B: Period 2) QIDS<11 Participants: Participants who were responders with QIDS-SR16 score <11 at the end of Period 1 continued to receive placebo intranasally (1 spray of placebo into each nostril at 0 and 5 minutes using 4 separate devices) on Days 8 and 11 in Period 2.
- Placebo to Esketamine 14mg (Panel B: Period 2): Participants who received placebo in Period 1 and were non-responders with QIDS-SR16 score >=11 at the end of Period 1 were re-randomized to receive esketamine 14 mg intranasally (1 spray of esketamine 14 mg into one nostril and 1 spray of placebo in other nostril at 0 minute and 1 spray of placebo in each nostril at 5 minutes using 4 separate devices) on Days 8 and 11 in Period 2.
- Placebo to Esketamine 56mg (Panel B: Period 2): Participants who received placebo in Period 1 and were non-responders (with QIDS-SR16 score >=11) at the end of Period 1 in Panel B were re-randomized to receive esketamine 56 mg intranasally (1 spray of esketamine 14 mg to each nostril at 0 and 5 minute and 1 spray of placebo to each nostril at 10 minutes) on Days 8 and 11 in Period 2.
- Esketamine 14 mg (Panel B: Period 2): Participants who received esketamine 14 mg in Period 1 of Panel B continued to receive esketamine 14 mg (1 spray of esketamine 14 mg to one nostril and 1 spray of placebo into other nostril at 0 minute and 1 spray of placebo to each nostril at 5 and 10 minutes) on Days 8 and 11 in Period 2.
- Esketamine 56 mg (Panel B: Period 2): Participants who received esketamine 56 mg in Period 1 of Panel B continued to receive esketamine 56 mg (1 spray of esketamine 14 mg to each nostril at 0 and 5 minute and 1 spray of placebo to each nostril at 10 minutes) on Days 8 and 11 in Period 2.
- Placebo/Placebo/Open Label Esketamine (Panel A): Participants who received Placebo in Period 1 and 2 of Panel A and elected to continue with open label phase received up to 9 single doses of intranasal esketamine on Days 15, 18, 22, 25, 32, 39, 46, 60 and 74. The doses for the optional open-label treatment phase included 28, 56, and 84 mg of esketamine. All participants started with intranasal esketamine 56 mg on Day 15. Subsequent doses on Days 18, 22, 25, 32, 39, and 46 could be adjusted to the next lower or higher dose, based on the investigator's clinical judgment. The same dose administered on Day 46 was administered on Day 60 and Day 74.
- Placebo/Esketamine/Open Label Esketamine (Panel A): Participants who received Placebo in Period 1 and esketamine in Period 2 of Panel A and elected to continue with open label phase received up to 9 single doses of intranasal esketamine on Days 15, 18, 22, 25, 32, 39, 46, 60 and 74. The doses for the optional open-label treatment phase included 28, 56, and 84 mg of esketamine. All participants started with intranasal esketamine 56 mg on Day 15. Subsequent doses on Days 18, 22, 25, 32, 39, and 46 could be adjusted to the next lower or higher dose, based on the investigator's clinical judgment. The same dose administered on Day 46 was administered on Day 60 and Day 74.
- Esketamine/Esketamine/Open Label Esketamine (Panel A): Participants who received esketamine in Period 1 and 2 of Panel A and elected to continue with open label phase received up to 9 single doses of intranasal esketamine on Days 15, 18, 22, 25, 32, 39, 46, 60 and 74. The doses for the optional open-label treatment phase included 28, 56, and 84 mg of esketamine. All participants started with intranasal esketamine 56 mg on Day 15. Subsequent doses on Days 18, 22, 25, 32, 39, and 46 could be adjusted to the next lower or higher dose, based on the investigator's clinical judgment. The same dose administered on Day 46 was administered on Day 60 and Day 74.
- Placebo/Placebo/Open Label Esketamine (Panel B): Participants who received Placebo in Period 1 and 2 of Panel A and elected to continue with open label phase received up to 4 single doses of intranasal esketamine on Days 15, 18, 22 and 25. The doses for the optional open-label treatment phase included 14, 28 and 56 mg of esketamine. All participants started with intranasal esketamine 56 mg on Day 15. Subsequent doses on Days 18, 22 and 25 could be adjusted to the next lower or higher dose, based on the investigator's clinical judgment.
- Placebo/Esketamine/Open Label Esketamine (Panel B): Participants who received Placebo in Period 1 and esketamine in Period 2 of Panel A and elected to continue with open label phase received up to 4 single doses of intranasal esketamine on Days 15, 18, 22 and 25. The doses for the optional open-label treatment phase included 14, 28 and 56 mg of esketamine. All participants started with intranasal esketamine 56 mg on Day 15. Subsequent doses on Days 18, 22 and 25 could be adjusted to the next lower or higher dose, based on the investigator's clinical judgment.
- Esketamine/Esketamine/Open Label Esketamine (Panel B): Participants who received esketamine in Period 1 and 2 of Panel A and elected to continue with open label phase received up to 4 single doses of intranasal esketamine on Days 15, 18, 22 and 25. The doses for the optional open-label treatment phase included 14, 28 and 56 mg of esketamine. All participants started with intranasal esketamine 56 mg on Day 15. Subsequent doses on Days 18, 22 and 25 could be adjusted to the next lower or higher dose, based on the investigator's clinical judgment.
- Placebo: Follow up Phase: All participants whose last dose was Placebo in the double-blind phase or open label phase and were not consent withdrawn were followed for safety for 8 weeks.
- Esketamine 14 mg: Follow up Phase: All participants whose last dose was esketamine 14 mg in the double-blind phase or open label phase and were not consent withdrawn were followed for safety for 8 weeks.
- Esketamine 28 mg: Follow up Phase: All participants whose last dose was esketamine 28 mg in the double-blind phase or open label phase and were not consent withdrawn were followed for safety for 8 weeks.
- Esketamine 56 mg: Follow up Phase: All participants whose last dose was esketamine 56 mg in the double-blind phase or open label phase and were not consent withdrawn were followed for safety for 8 weeks.
- Esketamine 84 mg: Follow up Phase: All participants whose last dose was esketamine 84 mg in the double-blind phase or open label phase and were not consent withdrawn were followed for safety for 8 weeks.
Period: Period 1 (Panel A and B)
Arm/Group | Placebo (Panel A: Period 1) | Esketamine 28 mg (Panel A: Period 1) | Esketamine 56 mg (Panel A: Period 1) | Esketamine 84 mg (Panel A: Period 1) | Placebo (Panel B: Period 1) | Esketamine 14 mg (Panel B: Period 1) | Esketamine 56 mg (Panel B: Period 1) | Placebo (Panel A: Period 2) QIDS >= 11 Participants | Placebo (Panel A: Period 2) QIDS<11 Participants | Placebo to Esketamine 28mg (Panel A: Period 2) | Placebo to Esketamine 56 mg (Panel A: Period 2) | Placebo to Esketamine 84 mg (Panel A: Period 2) | Esketamine 28 mg (Panel A: Period 2) | Esketamine 56 mg (Panel A: Period 2) | Esketamine 84 mg (Panel A: Period 2) | Placebo (Panel B: Period 2) QIDS >=11 Participants | Placebo (Panel B: Period 2) QIDS<11 Participants | Placebo to Esketamine 14mg (Panel B: Period 2) | Placebo to Esketamine 56mg (Panel B: Period 2) | Esketamine 14 mg (Panel B: Period 2) | Esketamine 56 mg (Panel B: Period 2) | Placebo/Placebo/Open Label Esketamine (Panel A) | Placebo/Esketamine/Open Label Esketamine (Panel A) | Esketamine/Esketamine/Open Label Esketamine (Panel A) | Placebo/Placebo/Open Label Esketamine (Panel B) | Placebo/Esketamine/Open Label Esketamine (Panel B) | Esketamine/Esketamine/Open Label Esketamine (Panel B) | Placebo: Follow up Phase | Esketamine 14 mg: Follow up Phase | Esketamine 28 mg: Follow up Phase | Esketamine 56 mg: Follow up Phase | Esketamine 84 mg: Follow up Phase
Started | 33 | 11 | 11 | 12 | 21 | 11 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rerandomized to Esketamine 56 mg | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rerandomized to Esketamine 28mg | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rerandomized to Esketamine 84mg | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 32 | 8 | 11 | 12 | 21 | 11 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 (Panel A and B)
Arm/Group | Placebo (Panel A: Period 1) | Esketamine 28 mg (Panel A: Period 1) | Esketamine 56 mg (Panel A: Period 1) | Esketamine 84 mg (Panel A: Period 1) | Placebo (Panel B: Period 1) | Esketamine 14 mg (Panel B: Period 1) | Esketamine 56 mg (Panel B: Period 1) | Placebo (Panel A: Period 2) QIDS >= 11 Participants | Placebo (Panel A: Period 2) QIDS<11 Participants | Placebo to Esketamine 28mg (Panel A: Period 2) | Placebo to Esketamine 56 mg (Panel A: Period 2) | Placebo to Esketamine 84 mg (Panel A: Period 2) | Esketamine 28 mg (Panel A: Period 2) | Esketamine 56 mg (Panel A: Period 2) | Esketamine 84 mg (Panel A: Period 2) | Placebo (Panel B: Period 2) QIDS >=11 Participants | Placebo (Panel B: Period 2) QIDS<11 Participants | Placebo to Esketamine 14mg (Panel B: Period 2) | Placebo to Esketamine 56mg (Panel B: Period 2) | Esketamine 14 mg (Panel B: Period 2) | Esketamine 56 mg (Panel B: Period 2) | Placebo/Placebo/Open Label Esketamine (Panel A) | Placebo/Esketamine/Open Label Esketamine (Panel A) | Esketamine/Esketamine/Open Label Esketamine (Panel A) | Placebo/Placebo/Open Label Esketamine (Panel B) | Placebo/Esketamine/Open Label Esketamine (Panel B) | Esketamine/Esketamine/Open Label Esketamine (Panel B) | Placebo: Follow up Phase | Esketamine 14 mg: Follow up Phase | Esketamine 28 mg: Follow up Phase | Esketamine 56 mg: Follow up Phase | Esketamine 84 mg: Follow up Phase
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 4 | 8 | 9 | 5 | 8 | 11 | 12 | 5 | 8 | 5 | 3 | 11 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 4 | 8 | 8 | 5 | 8 | 11 | 10 | 5 | 8 | 5 | 2 | 11 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open Label Phase (Optional)
Arm/Group | Placebo (Panel A: Period 1) | Esketamine 28 mg (Panel A: Period 1) | Esketamine 56 mg (Panel A: Period 1) | Esketamine 84 mg (Panel A: Period 1) | Placebo (Panel B: Period 1) | Esketamine 14 mg (Panel B: Period 1) | Esketamine 56 mg (Panel B: Period 1) | Placebo (Panel A: Period 2) QIDS >= 11 Participants | Placebo (Panel A: Period 2) QIDS<11 Participants | Placebo to Esketamine 28mg (Panel A: Period 2) | Placebo to Esketamine 56 mg (Panel A: Period 2) | Placebo to Esketamine 84 mg (Panel A: Period 2) | Esketamine 28 mg (Panel A: Period 2) | Esketamine 56 mg (Panel A: Period 2) | Esketamine 84 mg (Panel A: Period 2) | Placebo (Panel B: Period 2) QIDS >=11 Participants | Placebo (Panel B: Period 2) QIDS<11 Participants | Placebo to Esketamine 14mg (Panel B: Period 2) | Placebo to Esketamine 56mg (Panel B: Period 2) | Esketamine 14 mg (Panel B: Period 2) | Esketamine 56 mg (Panel B: Period 2) | Placebo/Placebo/Open Label Esketamine (Panel A) | Placebo/Esketamine/Open Label Esketamine (Panel A) | Esketamine/Esketamine/Open Label Esketamine (Panel A) | Placebo/Placebo/Open Label Esketamine (Panel B) | Placebo/Esketamine/Open Label Esketamine (Panel B) | Esketamine/Esketamine/Open Label Esketamine (Panel B) | Placebo: Follow up Phase | Esketamine 14 mg: Follow up Phase | Esketamine 28 mg: Follow up Phase | Esketamine 56 mg: Follow up Phase | Esketamine 84 mg: Follow up Phase
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 20 | 27 | 13 | 7 | 19 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 11 | 23 | 13 | 7 | 19 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 9 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Follow-up Phase
Arm/Group | Placebo (Panel A: Period 1) | Esketamine 28 mg (Panel A: Period 1) | Esketamine 56 mg (Panel A: Period 1) | Esketamine 84 mg (Panel A: Period 1) | Placebo (Panel B: Period 1) | Esketamine 14 mg (Panel B: Period 1) | Esketamine 56 mg (Panel B: Period 1) | Placebo (Panel A: Period 2) QIDS >= 11 Participants | Placebo (Panel A: Period 2) QIDS<11 Participants | Placebo to Esketamine 28mg (Panel A: Period 2) | Placebo to Esketamine 56 mg (Panel A: Period 2) | Placebo to Esketamine 84 mg (Panel A: Period 2) | Esketamine 28 mg (Panel A: Period 2) | Esketamine 56 mg (Panel A: Period 2) | Esketamine 84 mg (Panel A: Period 2) | Placebo (Panel B: Period 2) QIDS >=11 Participants | Placebo (Panel B: Period 2) QIDS<11 Participants | Placebo to Esketamine 14mg (Panel B: Period 2) | Placebo to Esketamine 56mg (Panel B: Period 2) | Esketamine 14 mg (Panel B: Period 2) | Esketamine 56 mg (Panel B: Period 2) | Placebo/Placebo/Open Label Esketamine (Panel A) | Placebo/Esketamine/Open Label Esketamine (Panel A) | Esketamine/Esketamine/Open Label Esketamine (Panel A) | Placebo/Placebo/Open Label Esketamine (Panel B) | Placebo/Esketamine/Open Label Esketamine (Panel B) | Esketamine/Esketamine/Open Label Esketamine (Panel B) | Placebo: Follow up Phase | Esketamine 14 mg: Follow up Phase | Esketamine 28 mg: Follow up Phase | Esketamine 56 mg: Follow up Phase | Esketamine 84 mg: Follow up Phase
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 12 | 39 | 42
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 12 | 39 | 42
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Panel A: Period 1) | Esketamine 28 mg (Panel A: Period 1) | Esketamine 56 mg (Panel A: Period 1) | Esketamine 84 mg (Panel A: Period 1) | Placebo (Panel B: Period 1) | Esketamine 14 mg (Panel B: Period 1) | Esketamine 56 mg (Panel B: Period 1) | Total
Number analyzed (Participants) | 33 | 11 | 11 | 12 | 21 | 11 | 9 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (9.60) | 42.1 (10.31) | 42.7 (11.23) | 49.8 (9.29) | 45.3 (7.66) | 42.2 (9.43) | 45.6 (7.35) | 44.6 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 5 | 9 | 6 | 9 | 4 | 4 | 55
  Male | 15 | 6 | 2 | 6 | 12 | 7 | 5 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 21 | 11 | 9 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 4 | 4 | 1 | 0 | 0 | 0 | 18
  White | 24 | 7 | 6 | 11 | 0 | 0 | 0 | 48
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Panel A and B: Change From Baseline (Day 1) in Montgomery Asberg Depression Rating Scale (MADRS) Total Score at Day 8- Analysis of Covariance (ANCOVA) Analysis
Description: MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition. A negative change in score indicates improvement.
Time Frame: Baseline (Day 1) and Endpoint (Day 8) of Period 1
Population: Period 1 Intent-to-treat (ITT) analysis set included all participants randomly assigned to treatment in period 1.
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Groups:
- Panel A: Period 1 Placebo: Participants self administered placebo intranasally (1 spray to each nostril at 0, 5 and 10 minutes) on Days 1 and 4 of Period 1.
- Panel A: Period 1 Esketamine 28 mg: Participants self administered esketamine 28 mg intranasally (1 spray of esketamine 14 mg to each nostril at 0 minute and 1 spray of placebo to each nostril at 5 and 10 minutes) on Days 1 and 4 of Period 1.
- Panel A: Period 1 Esketamine 56 mg: Participants self administered esketamine 56 mg intranasally (1 spray of esketamine 14 mg to each nostril at 0 and 5 minute and 1 spray of placebo to each nostril at 10 minutes) on Days 1 and 4 of Period 1.
- Panel A: Period 1 Esketamine 84 mg: Participants self administered esketamine 84 mg intranasally (1 spray of esketamine 14 mg to each nostril at 0, 5 and 10 minutes) on Days 1 and 4 of Period 1.
- Panel B: Period 1 Placebo: Participants self administered placebo intranasally (1 spray to each nostril at 0 and 5 minutes) on Days 1 and 4 of Period 1.
- Panel B: Period 1 Esketamine 14 mg: Participants self administered esketamine 14 mg intranasally (1 spray of esketamine 14 mg into one nostril and 1 spray of placebo into other nostril at 0 minute and then 1 spray of placebo to each nostril at 5 minutes) on Days 1 and 4 of Period 1.
- Panel B: Period 1 Esketamine 56 mg: Participants self administered esketamine 56 mg intranasally (1 spray of esketamine 14 mg into each nostril at 0 and 5 minutes) on Days 1 and 4 of Period 1.
Arm/Group | Panel A: Period 1 Placebo | Panel A: Period 1 Esketamine 28 mg | Panel A: Period 1 Esketamine 56 mg | Panel A: Period 1 Esketamine 84 mg | Panel B: Period 1 Placebo | Panel B: Period 1 Esketamine 14 mg | Panel B: Period 1 Esketamine 56 mg
Number analyzed (Participants) | 33 | 11 | 11 | 12 | 21 | 11 | 9
Unit on a scale | -4.9 (1.74) | -9.8 (2.72) | -12.4 (2.66) | -15.3 (2.56) | -6.6 (1.53) | -4.8 (2.13) | -10.3 (2.36)

2. Primary Outcome: Panel A and B: Change From Baseline (Day 8) in Montgomery Asberg Depression Rating Scale Total Score at Day 15- ANCOVA Analysis
Description: as for outcome 1
Time Frame: Baseline (Day 8) and Endpoint (Day 15) of Period 2
Population: Period 2 ITT analysis set included non-responders (QIDS-SR16 total score >=11) to placebo treatment in Period 1 and were then randomly re-assigned to a treatment group in Period 2. Only placebo participants with a QIDS-SR16 score >= 11 at End Point Period 1 who were re-randomized in Period 2 are included in the Period 2 summary.
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Groups:
- Panel A: Period 2 Placebo: Participants who were non-responders at the end of Period 1 in Panel A (with Quick Inventory of Depressive Symptomatology - 16-item Self Report (QIDS-SR16) score >=11) were randomly re-assigned to receive same Placebo (1 spray to each nostril at 0, 5 and 10 minutes) on Days 8 and 11 of Period 2.
- Panel A:Period 2 Esketamine 28 mg: Participants who were non-responders at the end of Period 1 in Panel A (with QIDS-SR 16 score >=11) were randomly re-assigned to receive esketamine 28 mg (1 spray of esketamine 14 mg to each nostril at 0 minute and 1 spray of placebo to each nostril at 5 and 10 minutes) on Days 8 and 11 of Period 2.
- Panel A: Period 2 Esketamine 56 mg: Participants who were non-responders at the end of Period 1 in Panel A (with QIDS-SR16 score >=11) were randomly re-assigned to receive esketamine 56 mg (1 spray of esketamine 14 mg to each nostril at 0 and 5 minute and 1 spray of placebo to each nostril at 10 minutes) on Days 8 and 11 of Period 2.
- Panel A: Period 2 Esketamine 84 mg: Participants who were non-responders at the end of Period 1 in Panel A (with QIDS-SR 16 score >=11) were randomly re-assigned to receive esketamine 84 mg (1 spray of esketamine 14 mg to each nostril at 0, 5 and 10 minutes) on Days 8 and 11 of Period 2.
- Panel B: Period 2 Placebo: Participants who were non-responders with QIDS-SR 16 score >=11 received placebo intranasally (1 spray of placebo into each nostril at 0 and 5 minutes) on Days 8 and 11 of Period 2.
- Panel B: Period 2 Esketamine 14 mg: Participants who received placebo in Period 1 and were non-responders with QIDS-SR16 score >=11 received esketamine 14 mg intranasally (1 spray of esketamine into one nostril and 1 spray of placebo in other nostril at 0 minutes and 1 spray of placebo in each nostril at 5 minutes) in Period 2.
- Panel B:Period 2 Esketamine 56 mg: Participants who were responders (with QIDS-SR16 score <11) at the end of Period 1 in Panel B continued to receive esketamine 56 mg (1 spray of esketamine 14 mg to each nostril at 0 and 5 minute and 1 spray of placebo to each nostril at 10 minutes) on Days 8 and 11 in Period 2.
Arm/Group | Panel A: Period 2 Placebo | Panel A:Period 2 Esketamine 28 mg | Panel A: Period 2 Esketamine 56 mg | Panel A: Period 2 Esketamine 84 mg | Panel B: Period 2 Placebo | Panel B: Period 2 Esketamine 14 mg | Panel B:Period 2 Esketamine 56 mg
Number analyzed (Participants) | 6 | 8 | 9 | 5 | 5 | 5 | 3
Unit on a scale | -4.5 (2.92) | -7.6 (2.49) | -8.9 (2.51) | -11.4 (2.68) | -0.7 (3.32) | -6.6 (4.02) | -1.2 (6.04)

3. Secondary Outcome: Panel A and B: Percentage of Participants With Sustained Response Based on MADRS Total Score in Participants Who Have Completed the Double-Blind Phase and Received the Same Treatment for Both Periods
Description: Sustained response was defined as at least 50% improvement from baseline in the MADRS total score with onset by Day 2 that is maintained to study Day 15. MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition.
Time Frame: Day 2 Up to Day 15
Population: Population analyzed included participants from double-blind (DB) ITT (who were randomly assigned to treatment during the double-blind phase) who completed the double-blind phase and received the same treatment for both periods.
Measure: Number; unit: Percentage of participants
Groups:
- Panel A: Placebo (Period 1 and 2): Participants who received same placebo (1 spray to each nostril at 0, 5 and 10 minutes) treatment in Period 1 and 2 of Panel A.
- Panel A: Esketamine 28 mg (Period 1 and 2): Participants who received same esketamine 28mg (1 spray of esketamine 14 mg to each nostril at 0 minute and 1 spray of placebo to each nostril at 5 and 10 minutes) treatment in Period 1 and 2 of Panel A.
- Panel A: Esketamine 56 mg (Period 1 and 2): Participants who received same esketamine 56 mg (1 spray of esketamine 14 mg to each nostril at 0 and 5 minute and 1 spray of placebo to each nostril at 10 minutes) treatment in Period 1 and 2 of Panel A.
- Panel A: Esketamine 84 mg (Period 1 and 2): Participants who received same esketamine 84 mg (1 spray of esketamine 14 mg to each nostril at 0, 5 and 10 minutes) treatment in Period 1 and 2 of Panel A.
- Panel B: Placebo (Period 1 and 2): Participants who received same placebo (1 spray to each nostril at 0 and 5 minutes) treatment in Period 1 and 2 of Panel B.
- Panel B: Esketamine 14 mg (Period 1 and 2): Participants who received same esketamine 14 mg (1 spray of esketamine 14 mg into one nostril and 1 spray of placebo into other nostril at 0 minute and then 1 spray of placebo to each nostril at 5 minutes) treatment in Period 1 and 2 of Panel B.
- Panel B: Esketamine 56 mg (Period 1 and 2): Participants who received same esketamine 56 mg (1 spray of esketamine 14 mg into each nostril at 0 and 5 minutes) treatment in Period 1 and 2 of Panel B.
Arm/Group | Panel A: Placebo (Period 1 and 2) | Panel A: Esketamine 28 mg (Period 1 and 2) | Panel A: Esketamine 56 mg (Period 1 and 2) | Panel A: Esketamine 84 mg (Period 1 and 2) | Panel B: Placebo (Period 1 and 2) | Panel B: Esketamine 14 mg (Period 1 and 2) | Panel B: Esketamine 56 mg (Period 1 and 2)
Number analyzed (Participants) | 10 | 8 | 11 | 10 | 13 | 11 | 9
Percentage of participants | 0 | 12.5 | 9.1 | 30.0 | 15.4 | 18.2 | 22.2

4. Secondary Outcome: Panel A and B: Percentage of Participants With Sustained Response Based on MADRS Total Score in Participants Who Received the Same Treatment for Both Periods, Including Participants Who Did Not Complete the Double-blind Phase
Description: Sustained response was defined as at least 50 percent (%) improvement from baseline in the MADRS total score with onset by Day 2 that is maintained to study Day 15. MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition.
Time Frame: Day 2 Up to Day 15
Population: Population analyzed included participants from DB ITT (who were randomly assigned to treatment during the double-blind phase) who received the same treatment for both periods, including participants who did not complete the double-blind Phase.
Measure: Number; unit: Percentage of participants
Arm/Group | Panel A: Placebo (Period 1 and 2) | Panel A: Esketamine 28 mg (Period 1 and 2) | Panel A: Esketamine 56 mg (Period 1 and 2) | Panel A: Esketamine 84 mg (Period 1 and 2) | Panel B: Placebo (Period 1 and 2) | Panel B: Esketamine 14 mg (Period 1 and 2) | Panel B: Esketamine 56 mg (Period 1 and 2)
Number analyzed (Participants) | 10 | 8 | 11 | 12 | 13 | 11 | 9
Percentage of participants | 0 | 12.5 | 9.1 | 25.0 | 15.4 | 18.2 | 22.2

5. Secondary Outcome: Panel A and B: Percentage of Participants With Response Based on MADRS Total Score
Description: A participant is defined a responder at a given time point if the percent improvement in MADRS is greater than or equal to (>=) 50%. Participant who do not meet such criterion, worsen or discontinue during the DB phase for any reason was considered as non-responders, that is, was assigned a value of 0. MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition.
Time Frame: Period 1: Days 1 (2 hour), 2 and 8 of Double-blind Phase
Population: Period 1 ITT analysis set included all participants randomly assigned to treatment in period 1.
Measure: Number; unit: Percentage of participants
Arm/Group | Panel A: Period 1 Placebo | Panel A: Period 1 Esketamine 28 mg | Panel A: Period 1 Esketamine 56 mg | Panel A: Period 1 Esketamine 84 mg | Panel B: Period 1 Placebo | Panel B: Period 1 Esketamine 14 mg | Panel B: Period 1 Esketamine 56 mg
Number analyzed (Participants) | 33 | 11 | 11 | 12 | 21 | 11 | 9
Percentage of participants
  Day 1 (2 hour) | 18.2 | 54.5 | 36.4 | 58.3 | 33.3 | 36.4 | 44.4
  Day 2 | 3.0 | 36.4 | 27.3 | 41.7 | 28.6 | 36.4 | 44.4
  Day 8 | 6.1 | 9.1 | 18.2 | 41.7 | 23.8 | 18.2 | 22.2

6. Secondary Outcome: Panel A and B: Percentage of Participants With Response Based on MADRS Total Score
Description: A participant is defined a responder at a given time point if the percent improvement in MADRS is >=50%. Participant who do not meet such criterion, worsen or discontinue during the DB phase for any reason was considered as non-responders, that is, was assigned a value of 0. MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition.
Time Frame: Period 2: Days 1 (2 hour), 2 and 8 of Double-blind Phase
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Groups:
- Panel A: Period 2 Esketamine 28 mg: Participants who were non-responders at the end of Period 1 in Panel A (with QIDS-SR 16 score >=11) were randomly re-assigned to receive esketamine 28 mg (1 spray of esketamine 14 mg to each nostril at 0 minute and 1 spray of placebo to each nostril at 5 and 10 minutes) on Days 8 and 11 of Period 2.
- Panel B: Period 2 Esketamine 56 mg: Participants who were responders (with QIDS-SR16 score <11) at the end of Period 1 in Panel B continued to receive esketamine 56 mg (1 spray of esketamine 14 mg to each nostril at 0 and 5 minute and 1 spray of placebo to each nostril at 10 minutes) on Days 8 and 11 in Period 2.
Arm/Group | Panel A: Period 2 Placebo | Panel A: Period 2 Esketamine 28 mg | Panel A: Period 2 Esketamine 56 mg | Panel A: Period 2 Esketamine 84 mg | Panel B: Period 2 Placebo | Panel B: Period 2 Esketamine 14 mg | Panel B: Period 2 Esketamine 56 mg
Number analyzed (Participants) | 6 | 8 | 9 | 5 | 5 | 5 | 3
Percentage of participants
  Day 1 (2 hour) | 16.7 | 12.5 | 22.2 | 40.0 | 0 | 60.0 | 0
  Day 2 | 0 | 0 | 11.1 | 40.0 | 0 | 80.0 | 0
  Day 8 | 0 | 12.5 | 0 | 20.0 | 0 | 0 | 33.3

7. Secondary Outcome: Panel A and B: Percentage of Participants in Remission Based on MADRS Total Score at Days 1, 2 and 8 of Double-blind Phase
Description: Participants who had a MADRS total score of <=10 were considered remitters. MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition.
Time Frame: Days 1, 2 and 8 of Double-blind Phase of Period 1
Population: Period 1 ITT analysis set included all participants randomly assigned to treatment in period 1.
Measure: Number; unit: Percentage of participants
Groups:
- Panel A: Period 1: Placebo: Participants self administered placebo intranasally (1 spray to each nostril at 0, 5 and 10 minutes) on Days 1 and 4 of Period 1.
- Panel A: Period 1: Esketamine 56 mg: Participants self administered esketamine 56 mg intranasally (1 spray of esketamine 14 mg to each nostril at 0 and 5 minute and 1 spray of placebo to each nostril at 10 minutes) on Days 1 and 4 of Period 1.
Arm/Group | Panel A: Period 1: Placebo | Panel A: Period 1 Esketamine 28 mg | Panel A: Period 1: Esketamine 56 mg | Panel A: Period 1 Esketamine 84 mg | Panel B: Period 1 Placebo | Panel B: Period 1 Esketamine 14 mg | Panel B: Period 1 Esketamine 56 mg
Number analyzed (Participants) | 33 | 11 | 11 | 12 | 21 | 11 | 9
Percentage of participants
  Day 1 | 3.0 | 27.3 | 18.2 | 25.0 | 19.0 | 36.4 | 33.3
  Day 2 | 0 | 36.4 | 18.2 | 25.0 | 19.0 | 27.3 | 33.3
  Day 8 | 3.0 | 9.1 | 9.1 | 25.0 | 14.3 | 18.2 | 22.2

8. Secondary Outcome: Panel A and B: Percentage of Participants in Remission Based on MADRS Total Score at Days 1, 2 and 8 of Double-blind Phase
Description: Participants who had a MADRS total score of less than or equal to (<=10) were considered remitters. MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition. A negative change in score indicates improvement.
Time Frame: Days 1, 2 and 8 of Double-blind Phase of Period 2
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Panel A: Period 2 Placebo | Panel A: Period 2 Esketamine 28 mg | Panel A: Period 2 Esketamine 56 mg | Panel A: Period 2 Esketamine 84 mg | Panel B: Period 2 Placebo | Panel B: Period 2 Esketamine 14 mg | Panel B: Period 2 Esketamine 56 mg
Number analyzed (Participants) | 6 | 8 | 9 | 5 | 5 | 5 | 3
Percentage of participants
  Day 1 | 16.7 | 12.5 | 0 | 40.0 | 0 | 60.0 | 0
  Day 2 | 0 | 0 | 0 | 20.0 | 0 | 80.0 | 0
  Day 8 | 0 | 12.5 | 0 | 20.0 | 0 | 0 | 0

9. Secondary Outcome: Panel A and B: Change From Baseline (Day 1) in Quick Inventory of Depressive Symptomatology-16-item Self Report (QIDS-SR16) Total Score at Day 8 in the Double-Blind Treatment Phase- ANCOVA Analysis
Description: QIDS-SR16 is self-rated scale assesses severity of depressive symptoms. Total scores range from 0-27. Higher score indicates greater severity of depression. Negative change in score indicates improvement. Total score obtained by adding scores for each of 9 symptom domains of Diagnostic and Statistical Manual of Mental Disorders-4th edition major depressive disorder (DSM-IV MDD) criteria: depressed mood, loss of interest/pleasure, concentration/decision making, self-outlook, suicidal ideation, energy/fatigability, sleep, weight/appetite change, psychomotor changes. 16 items used to rate 9 criterion domains: 4 items used to rate sleep disturbance (early/middle/late insomnia/hypersomnia); 2 items used to rate psychomotor disturbance (agitation, retardation); 4 items used to rate appetite/weight disturbance. 1 item used to rate 6 domains (depressed mood, decreased interest, decreased energy, worthlessness/guilt, concentration/decision making, suicidal ideation). Each item was rated 0-3.
Time Frame: Baseline (Day 1) and Endpoint (Day 8) of Period 1
Population: Period 1 ITT analysis set included all participants randomly assigned to treatment in period 1.
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Panel A: Period 1 Placebo | Panel A: Period 1 Esketamine 28 mg | Panel A: Period 1 Esketamine 56 mg | Panel A: Period 1 Esketamine 84 mg | Panel B: Period 1 Placebo | Panel B: Period 1 Esketamine 14 mg | Panel B: Period 1 Esketamine 56 mg
Number analyzed (Participants) | 33 | 11 | 11 | 12 | 21 | 11 | 9
Unit on a scale | -1.8 (0.93) | -4.0 (1.43) | -4.4 (1.43) | -4.2 (1.39) | -1.1 (0.78) | -0.6 (1.10) | -3.0 (1.20)

10. Secondary Outcome: Panel A and B: Change From Baseline (Day 8) in Quick Inventory of Depressive Symptomatology-16-item Self Report Total Score at Day 15 in the Double-Blind Treatment Phase- ANCOVA Analysis
Description: as for outcome 9
Time Frame: Baseline (Day 8) and Endpoint (Day 15) of Period 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Panel A: Period 2 Placebo | Panel A: Period 2 Esketamine 28 mg | Panel A: Period 2 Esketamine 56 mg | Panel A: Period 2 Esketamine 84 mg | Panel B: Period 2 Placebo | Panel B: Period 2 Esketamine 14 mg | Panel B: Period 2 Esketamine 56 mg
Number analyzed (Participants) | 6 | 8 | 9 | 5 | 5 | 5 | 3
Unit on a scale | -2.0 (1.50) | -3.1 (1.35) | -2.0 (1.41) | -3.3 (1.48) | -2.1 (1.78) | -5.7 (1.78) | -1.5 (2.31)

11. Secondary Outcome: Panel A and B: Change From Baseline (Day 1) in Clinical Global Impression - Severity (CGI-S) Total Score at Day 8 in the Double-Blind Treatment Phase- ANCOVA Analysis on Ranks
Description: CGI-S provides measure of severity of participant's illness including participant's history, psychosocial circumstances, symptoms, behavior and impact of symptoms on ability to function. CGI-S evaluates severity of psychopathology on scale of 0 to 7. Considering total clinical experience, participant is assessed on severity of mental illness according to: 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among most extremely ill patients. CGI-S permits global evaluation of participant's condition at given time. A negative change in score indicates improvement.
Time Frame: Baseline (Day 1) and Endpoint (Day 8) of Period 1
Population: Period 1 ITT analysis set included all participants randomly assigned to treatment in period 1.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Panel A: Period 1 Placebo | Panel A: Period 1 Esketamine 28 mg | Panel A: Period 1 Esketamine 56 mg | Panel A: Period 1 Esketamine 84 mg | Panel B: Period 1 Placebo | Panel B: Period 1 Esketamine 14 mg | Panel B: Period 1 Esketamine 56 mg
Number analyzed (Participants) | 33 | 11 | 11 | 12 | 21 | 11 | 9
Units on a scale | 5.0 [1 to 6] | 4.0 [3 to 5] | 4.0 [1 to 5] | 4.0 [1 to 6] | 4.0 [1 to 6] | 4.0 [2 to 6] | 3.0 [3 to 6]

12. Secondary Outcome: Panel A and B: Change From Baseline (Day 8) in Clinical Global Impression - Severity Total Score at Day 15 in the Double-Blind Treatment Phase- ANCOVA Analysis on Ranks
Description: as for outcome 11
Time Frame: Baseline (Day 8) and Endpoint (Day 15) of Period 2
Population: as for outcome 2
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Panel A: Period 2 Placebo | Panel A: Period 2 Esketamine 28 mg | Panel A: Period 2 Esketamine 56 mg | Panel A: Period 2 Esketamine 84 mg | Panel B: Period 2 Placebo | Panel B: Period 2 Esketamine 14 mg | Panel B: Period 2 Esketamine 56 mg
Number analyzed (Participants) | 6 | 8 | 9 | 5 | 5 | 5 | 3
Units on a scale | 5.0 [4 to 5] | 4.0 [3 to 5] | 5.0 [4 to 6] | 4.0 [3 to 5] | 4.0 [3 to 6] | 3.0 [3 to 4] | 4.0 [4 to 5]

13. Secondary Outcome: Panel A and B: Change From Baseline (Day 1) in Generalized Anxiety Disorder (GAD-7) Total Score at Day 8 (Double-Blind Treatment Phase) ANCOVA Analysis
Description: GAD-7 is a brief and validated 7-item self-report assessment of overall anxiety. Participants respond to each item using a 4-point scale with response categories of 0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day. Item responses are summed to yield a total score with a range of 0 to 21, where higher scores indicate more anxiety. The recall period is 2 weeks. The severity of the GAD-7 is categorized as follows: None (0-4), Mild (5-9), Moderate (10-14) and Severe (15 -21).
Time Frame: Baseline (Day 1) and Endpoint (Day 8) of Period 1
Population: Period 1 ITT analysis set included all participants randomly assigned to treatment in period 1.
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Panel A: Period 1 Placebo | Panel A: Period 1 Esketamine 28 mg | Panel A: Period 1 Esketamine 56 mg | Panel A: Period 1 Esketamine 84 mg | Panel B: Period 1 Placebo | Panel B: Period 1 Esketamine 14 mg | Panel B: Period 1 Esketamine 56 mg
Number analyzed (Participants) | 33 | 11 | 11 | 12 | 21 | 11 | 9
Unit on a scale | -1.7 (0.88) | -1.5 (1.34) | -3.1 (1.34) | -5.1 (1.30) | -1.7 (0.68) | -1.9 (0.94) | -3.2 (1.03)

14. Secondary Outcome: Panel A and B: Change From Baseline (Day 8) in Generalized Anxiety Disorder-7 Total Score at Day 15 (Double-Blind Treatment Phase)- ANCOVA Analysis
Description: as for outcome 13
Time Frame: Baseline (Day 8) and Endpoint (Day 15) of Period 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Panel A: Period 2 Placebo | Panel A: Period 2 Esketamine 28 mg | Panel A: Period 2 Esketamine 56 mg | Panel A: Period 2 Esketamine 84 mg | Panel B: Period 2 Placebo | Panel B: Period 2 Esketamine 14 mg | Panel B: Period 2 Esketamine 56 mg
Number analyzed (Participants) | 6 | 8 | 9 | 5 | 5 | 5 | 3
Unit on a scale | 0.4 (1.02) | -1.6 (0.87) | 1.0 (0.98) | -0.9 (1.02) | -2.7 (1.68) | -6.6 (1.68) | -0.7 (2.27)

15. Secondary Outcome: Panel A and B: Change From Baseline (Day 1) in Patient Global Impression of Severity (PGI-S) Score Total Score at Day 8 in the Double-Blind Treatment Phase- ANCOVA Analysis on Ranks
Description: PGI-S is a patient-rated scale that assesses the severity of their illness at the time of assessment, relative to participants past experience. It is a 4-point (1 to 4) scale in response to the question 'Considering all aspects of your depression right now would you say your depression is?' with scores as follows: 1: none; 2: mild; 3: moderate; 4: severe. A higher score implies a more severe condition.
Time Frame: Baseline (Day 1) and Endpoint (Day 8) of Period 1
Population: Period 1 ITT analysis set included all participants randomly assigned to treatment in period 1.
Measure: Median (Full Range); unit: Unit on a scale
Arm/Group | Panel A: Period 1 Placebo | Panel A: Period 1 Esketamine 28 mg | Panel A: Period 1 Esketamine 56 mg | Panel A: Period 1 Esketamine 84 mg | Panel B: Period 1 Placebo | Panel B: Period 1 Esketamine 14 mg | Panel B: Period 1 Esketamine 56 mg
Number analyzed (Participants) | 33 | 11 | 11 | 12 | 21 | 11 | 9
Unit on a scale | 3.0 [2 to 4] | 3.0 [1 to 4] | 3.0 [1 to 3] | 3.0 [1 to 4] | 3.0 [2 to 4] | 3.0 [1 to 3] | 3.0 [2 to 3]

16. Secondary Outcome: Panel A and B: Change From Baseline (Day 8) in Patient Global Impression of Severity Score Total Score at Day 15 in the Double-Blind Treatment Phase- ANCOVA Analysis on Ranks
Description: PGI-S is a patient-rated scale that assesses the severity of their illness at the time of assessment, relative to participants past experience. It is a 4-point (1 to 4) scale in response to the question 'Considering all aspects of your depression right now would you say your depression is?' with scores as follows: 1: none; 2: mild; 3: moderate; 4: severe. A higher score implies a more severe condition. A negative change in score indicates improvement.
Time Frame: Baseline (Day 8) and Endpoint (Day 15) of Period 2
Population: as for outcome 2
Measure: Median (Full Range); unit: Unit on a scale
Arm/Group | Panel A: Period 2 Placebo | Panel A: Period 2 Esketamine 28 mg | Panel A: Period 2 Esketamine 56 mg | Panel A: Period 2 Esketamine 84 mg | Panel B: Period 2 Placebo | Panel B: Period 2 Esketamine 14 mg | Panel B: Period 2 Esketamine 56 mg
Number analyzed (Participants) | 6 | 8 | 9 | 5 | 5 | 5 | 3
Unit on a scale | 3.0 [2 to 4] | 3.0 [2 to 4] | 4.0 [2 to 4] | 3.0 [2 to 4] | 3.0 [2 to 3] | 3.0 [2 to 3] | 3.0 [2 to 4]

ADVERSE EVENTS:
Time Frame: Up to 21 weeks
Description: Safety analysis set for double-blind and open-label phase included all randomized participants who receive at least 1 dose of study drug in the respective phases. For follow-up phase safety population included all participants who entered in follow up phase.
Groups:
- Placebo (Panel A and B: Period 1): Panel A: Participants self-administered placebo intranasally (1 spray to each nostril at 0, 5 and 10 minutes) on Days 1 and 4 of Period 1 in Panel A. Panel B: Participants self-administered placebo intranasally (1 spray to each nostril at 0 and 5 minutes) on Days 1 and 4 of Period 1 in Panel B.
- Placebo (Panel A and B: Period 2) QIDS >=11 Participants: Panel A: Participants who were non-responders at the end of Period 1 in Panel A (with QIDS-SR16 score >=11) were randomly reassigned to receive same Placebo (1 spray to each nostril at 0, 5 and 10 minutes) on Days 8 and 11 of Period 2 in Panel A. Panel B: Participants who were non-responders with QIDS-SR16 score >=11 at the end of Period 1 were randomly assigned to receive placebo intranasally (1 spray of placebo into each nostril at 0 and 5 minutes using 4 separate devices) on Days 8 and 11 of Period 2 in Panel B.
- Placebo to Esketamine 14mg (Panel B: Period 2): Participants who received placebo in Period 1 and were non-responders with QIDS-SR16 score >=11 at the end of Period 1 were randomly reassigned to receive esketamine 14 mg intranasally (1 spray of esketamine 14 mg into once nostril and 1 spray of placebo in other nostril at 0 minute and 1 spray of placebo in each nostril at 5 minutes using 4 separate devices) on Days 8 and 11 in Period 2 of Panel B.
- Placebo to Esketamine 28mg (Panel A: Period 2): Participants who were non-responders at the end of Period 1 in Panel A (with QIDS-SR16 score >=11) were randomly reassigned to receive esketamine 28 mg (1 spray of esketamine 14 mg to each nostril at 0 minute and 1 spray of placebo to each nostril at 5 and 10 minutes) on Days 8 and 11 of Period 2 in Panel A.
- Placebo to Esketamine 56mg (Panel A and B: Period 2): Panel A: Participants who were non-responders at the end of Period 1 in Panel A (with QIDS-SR16 score >=11) were randomly reassigned to receive esketamine 56 mg (1 spray of esketamine 14 mg to each nostril at 0 and 5 minute and 1 spray of placebo to each nostril at 10 minutes) on Days 8 and 11 of Period 2 in Panel A. Panel B: Participants who were responders (with QIDS-SR16 score <11) at the end of Period 1 in Panel B continued to receive esketamine 56 mg (1 spray of esketamine 14 mg to each nostril at 0 and 5 minute and 1 spray of placebo to each nostril at 10 minutes) on Days 8 and 11 in Period 2 of Panel B.
- Placebo to Esketamine 84 mg (Panel A: Period 2): Participants who were non-responders at the end of Period 1 in Panel A (with QIDS-SR16 score >=11) were randomly reassigned to receive esketamine 84 mg (1 spray of esketamine 14 mg to each nostril at 0, 5 and 10 minutes) on Days 8 and 11 of Period 2 in Panel A.
- Placebo (Panel A and Panel B: Period 2): All participants who received placebo in Period 2 of Panel A and B (including participants with QIDS-SR16 score >=11 and QIDS-SR16 score <11) in double-blind phase.
- Esketamine 14 mg (Panel B: Period 2): Participants who received esketamine 14 mg in Period 1 of Panel B continued to receive esketamine 14 mg (1 spray of esketamine 14 mg to each nostril at 0 and 5 minute and 1 spray of placebo to each nostril at 10 minutes) on Days 8 and 11 in Period 2 of Panel B.
- Esketamine 28 mg (Panel A: Period 2): Participants who received esketamine 28 mg in Period 1 of Panel A continued to receive esketamine 28 mg (1 spray of esketamine 14 mg to each nostril at 0 minute and 1 spray of placebo to each nostril at 5 and 10 minutes) on Days 8 and 11 of Period 2 in Panel A.
- Esketamine 56 mg (Panel A and B: Period 2): Panel A: Participants who were non-responders at the end of Period 1 in Panel A (with QIDS-SR16 score >=11) were randomly re-assigned to receive esketamine 56 mg (1 spray of esketamine 14 mg to each nostril at 0 and 5 minute and 1 spray of placebo to each nostril at 10 minutes) on Days 8 and 11 of Period 2. Panel B: Participants who were responders (with QIDS-SR16 score <11) at the end of Period 1 in Panel B continued to receive esketamine 56 mg (1 spray of esketamine 14 mg to each nostril at 0 and 5 minute and 1 spray of placebo to each nostril at 10 minutes) on Days 8 and 11 in Period 2.
- Placebo/Placebo/Open Label Esketamine (Panel A and B): Panel A: Participants who received Placebo in Period 1 and 2 of Panel A and elected to continue with open label (OL) phase received up to 9 single doses of intranasal esketamine on Days 15,18,22,25,32, 39, 46,60,74. Doses for optional OL phase included 28, 56, and 84 mg of esketamine. All participants started with intranasal esketamine 56 mg on Day 15. Subsequent doses on Days 18,22,25,32,39,46 could be adjusted to next lower or higher dose, based on investigator's clinical judgment. Same dose administered on Day 46 was administered on Day 60, 74. Panel B: Participants who received Placebo in Period 1 and 2 of Panel A and elected to continue with OL phase received up to 4 single doses of intranasal esketamine on Days 15, 18, 22, 25. Doses for OL phase included 14, 28, 56 mg of esketamine. All participants started with intranasal esketamine 56 mg on Day 15. Subsequent doses on Days 18, 22, 25 could be adjusted to next lower or higher dose, based on investigator's clinical judgment.
- Placebo/Esketamine/Open Label Esketamine (Panel A and B): Panel A: Participants who received Placebo in Period 1, esketamine in Period 2 and elected to continue with OL phase received up to 9 single doses of intranasal esketamine on Days 15,18,22,25,32,39,46,60, 74. Doses for OL phase included 28,56,84 mg of esketamine. All participants started with intranasal esketamine 56 mg on Day 15. Subsequent doses on Days 18,22,25,32,39, 46 could be adjusted to the next lower or higher dose, based on the investigator's clinical judgment. Same dose administered on Day 46 was administered on Day 60,74. Panel B: Participants who received Placebo in Period 1 and esketamine in Period 2 of Panel A and elected to continue with OL phase received up to 4 single doses of intranasal esketamine on Days 15,18,22,25. Doses for OL phase included 14,28,56 mg of esketamine. All participants started with intranasal esketamine 56 mg on Day 15. Subsequent doses on Days 18,22,25 could be adjusted to next lower or higher dose, based on the investigator's clinical judgment.
- Esketamine/Esketamine/Open Label Esketamine (Panel A and B): Panel A: Participants who received esketamine in Period 1 and 2 and elected to continue with open label phase received up to 9 single doses of intranasal esketamine on Days 15,18,22,25,32,39,46,60,74. Doses for OL treatment phase included 28, 56, 84 mg of esketamine. All participants started with intranasal esketamine 56 mg on Day 15. Subsequent doses on Days 18, 22,25,32,39, 46 could be adjusted to the next lower or higher dose, based on the investigator's clinical judgment. Same dose administered on Day 46 was administered on Day 60,74.Panel B: Participants who received esketamine in Period 1 and 2 of Panel A and elected to continue with OL phase received up to 4 single doses of intranasal esketamine on Days 15, 18, 22, 25. Doses for OL phase included 14, 28, 56 mg of esketamine. All participants started with intranasal esketamine 56 mg on Day 15. Subsequent doses on Days 18, 22, 25 could be adjusted to the next lower or higher dose, based on the investigator's clinical judgment.
- Esketamine 56 mg (Panel A and B: Period 1): Panel A: Participants self administered esketamine 56 mg intranasally (1 spray of esketamine 14 mg to each nostril at 0 and 5 minute and 1 spray of placebo to each nostril at 10 minutes) on Days 1 and 4 of Period 1. Panel B: Participants self administered esketamine 56 mg intranasally (1 spray of esketamine 14 mg into each nostril at 0 and 5 minutes) on Days 1 and 4 of Period 1.
- Esketamine 84 mg (Panel A: Period 2): Participants who received esketamine 84 mg in Period 1 of Panel A continued to receive esketamine 84 mg (1 spray of esketamine 14 mg to each nostril at 0, 5 and 10 minutes) on Days 8 and 11 of Period 2 in Panel A.
Arm/Group | Placebo (Panel A and B: Period 1) | Esketamine 28 mg (Panel A: Period 1) | Placebo (Panel A and B: Period 2) QIDS >=11 Participants | Placebo to Esketamine 14mg (Panel B: Period 2) | Placebo to Esketamine 28mg (Panel A: Period 2) | Placebo to Esketamine 56mg (Panel A and B: Period 2) | Placebo to Esketamine 84 mg (Panel A: Period 2) | Placebo (Panel A and Panel B: Period 2) | Esketamine 14 mg (Panel B: Period 2) | Esketamine 28 mg (Panel A: Period 2) | Esketamine 56 mg (Panel A and B: Period 2) | Placebo/Placebo/Open Label Esketamine (Panel A and B) | Placebo/Esketamine/Open Label Esketamine (Panel A and B) | Esketamine/Esketamine/Open Label Esketamine (Panel A and B) | Placebo: Follow up Phase | Esketamine 14 mg: Follow up Phase | Esketamine 28 mg: Follow up Phase | Esketamine 56 mg: Follow up Phase | Esketamine 84 mg: Follow up Phase | Esketamine 14 mg (Panel B: Period 1) | Esketamine 56 mg (Panel A and B: Period 1) | Esketamine 84 mg (Panel A: Period 1) | Esketamine 84 mg (Panel A: Period 2)
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/11 | 1/23 | 0/5 | 0/8 | 0/12 | 0/5 | 1/23 | 0/16 | 0/16 | 0/32 | 0/23 | 0/27 | 1/46 | 0/1 | 0/4 | 1/12 | 1/39 | 1/42 | 0/11 | 0/20 | 0/12 | 0/17
Other Adverse Events (participants affected / at risk) | 27/54 | 8/11 | 15/23 | 5/5 | 4/8 | 11/12 | 5/5 | 12/23 | 11/16 | 8/16 | 26/32 | 23/23 | 22/27 | 39/46 | 0/1 | 1/4 | 4/12 | 10/39 | 7/42 | 6/11 | 18/20 | 10/12 | 12/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (Panel A and B: Period 1) (N=54) | Esketamine 28 mg (Panel A: Period 1) (N=11) | Placebo (Panel A and B: Period 2) QIDS >=11 Participants (N=23) | Placebo to Esketamine 14mg (Panel B: Period 2) (N=5) | Placebo to Esketamine 28mg (Panel A: Period 2) (N=8) | Placebo to Esketamine 56mg (Panel A and B: Period 2) (N=12) | Placebo to Esketamine 84 mg (Panel A: Period 2) (N=5) | Placebo (Panel A and Panel B: Period 2) (N=23) | Esketamine 14 mg (Panel B: Period 2) (N=16) | Esketamine 28 mg (Panel A: Period 2) (N=16) | Esketamine 56 mg (Panel A and B: Period 2) (N=32) | Placebo/Placebo/Open Label Esketamine (Panel A and B) (N=23) | Placebo/Esketamine/Open Label Esketamine (Panel A and B) (N=27) | Esketamine/Esketamine/Open Label Esketamine (Panel A and B) (N=46) | Placebo: Follow up Phase (N=1) | Esketamine 14 mg: Follow up Phase (N=4) | Esketamine 28 mg: Follow up Phase (N=12) | Esketamine 56 mg: Follow up Phase (N=39) | Esketamine 84 mg: Follow up Phase (N=42) | Esketamine 14 mg (Panel B: Period 1) (N=11) | Esketamine 56 mg (Panel A and B: Period 1) (N=20) | Esketamine 84 mg (Panel A: Period 1) (N=12) | Esketamine 84 mg (Panel A: Period 2) (N=17)
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General Physical Health Deterioration (General disorders) | 0/1 | 0/3 | 0 | 0 | 0 | 0 | 0 | 0/11 | 0/8 | 0 | 0/12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/1 | 0/3 | 0 | 0 | 0 | 0 | 0 | 0/11 | 0/8 | 0 | 0/12 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA
Completed Suicide (Psychiatric disorders) | 0/1 | 0/3 | 0 | 0 | 0 | 0 | 0 | 0/11 | 0/8 | 0 | 0/12 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA
Confusional State (Psychiatric disorders) | 0/1 | 0/3 | 0 | 0 | 0 | 0 | 0 | 0/11 | 0/8 | 0 | 0/12 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (Panel A and B: Period 1) (N=54) | Esketamine 28 mg (Panel A: Period 1) (N=11) | Placebo (Panel A and B: Period 2) QIDS >=11 Participants (N=23) | Placebo to Esketamine 14mg (Panel B: Period 2) (N=5) | Placebo to Esketamine 28mg (Panel A: Period 2) (N=8) | Placebo to Esketamine 56mg (Panel A and B: Period 2) (N=12) | Placebo to Esketamine 84 mg (Panel A: Period 2) (N=5) | Placebo (Panel A and Panel B: Period 2) (N=23) | Esketamine 14 mg (Panel B: Period 2) (N=16) | Esketamine 28 mg (Panel A: Period 2) (N=16) | Esketamine 56 mg (Panel A and B: Period 2) (N=32) | Placebo/Placebo/Open Label Esketamine (Panel A and B) (N=23) | Placebo/Esketamine/Open Label Esketamine (Panel A and B) (N=27) | Esketamine/Esketamine/Open Label Esketamine (Panel A and B) (N=46) | Placebo: Follow up Phase (N=1) | Esketamine 14 mg: Follow up Phase (N=4) | Esketamine 28 mg: Follow up Phase (N=12) | Esketamine 56 mg: Follow up Phase (N=39) | Esketamine 84 mg: Follow up Phase (N=42) | Esketamine 14 mg (Panel B: Period 1) (N=11) | Esketamine 56 mg (Panel A and B: Period 1) (N=20) | Esketamine 84 mg (Panel A: Period 1) (N=12) | Esketamine 84 mg (Panel A: Period 2) (N=17)
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear Congestion (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 2 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Accommodation Disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival Hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Visual Impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 3 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2
Nausea (Gastrointestinal disorders) | 5 | 2 | 3 | 1 | 0 | 2 | 2 | 2 | 1 | 1 | 3 | 4 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 2 | 2
Oral Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia Oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Salivary Hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Energy Increased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feeling Abnormal (General disorders) | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 1 | 4 | 0 | 3 | 4 | 4 | 7 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 1 | 1
Feeling Drunk (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling Hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling Jittery (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait Disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hangover (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Product Taste Abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Sluggishness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 5 | 1 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood Pressure Diastolic Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood Pressure Increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 4 | 3 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1
Blood Pressure Systolic Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oxygen Saturation Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Altered State of Consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coordination Abnormal (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in Attention (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 4 | 0 | 2 | 0 | 4 | 3 | 0 | 2 | 2 | 11 | 7 | 9 | 14 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 5 | 5
Dizziness Postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 9 | 2 | 6 | 1 | 1 | 2 | 3 | 4 | 2 | 1 | 4 | 4 | 6 | 9 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 4
Dysgraphia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 4 | 5 | 0 | 2 | 3 | 1 | 4 | 1 | 2 | 3 | 4 | 5 | 5 | 0 | 1 | 0 | 0 | 4 | 2 | 4 | 2 | 1
Hypersomnia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 3 | 0 | 4 | 3 | 4 | 8 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0
Loss of Consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental Impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Psychomotor Hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1
Slow Speech (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 3 | 1 | 7 | 1 | 0 | 2 | 0 | 6 | 1 | 1 | 5 | 7 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tunnel Vision (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Visual Field Defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Daydreaming (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dissociation (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 4 | 1 | 0 | 1 | 0 | 8 | 2 | 4 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 2
Dissociative Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 4 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3
Dysphoria (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fear (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination, Visual (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Illusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Merycism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somatic Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suspiciousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thinking Abnormal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bladder Pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Micturition Urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nasal Mucosal Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal Pruritus (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Pharyngeal Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal Hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Peripheral Coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0/1 | 0/3 | 0 | 0 | 0 | 0 | 0 | 0/11 | 0/8 | 0 | 0/12 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis Allergic (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0/12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erosive Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/32 | 0 | 0 | 0 | 0 | 0
Oesophageal Stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
C-Reactive Protein Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sensory Disturbance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depersonalisation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Persecutory Delusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.